CLINICAL TRIAL: NCT04969133
Title: TAP Block Versus Local Anesthesia Infiltration at Wound Site for Postoperative Pain Relief After Laparoscopic Appendicectomy in Children
Brief Title: TAP Block Versus Local Anesthesia Wound Infiltration for Postoperative Pain Relief After Appendicectomy in Children
Acronym: PABLO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2021/571
Record Dates: First submitted 2021-06-18; First posted 2021-07-20 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-01

CONDITIONS: Appendicitis Acute; Pediatrics; Analgesia
Keywords: Appendicectomy; Laparoscopy; infiltration; TAP block
MeSH Terms: conditions — Appendicitis; Agnosia | interventions — Levobupivacaine

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP Block (Active Comparator): Transverse abdominal block is realisated at the beginning of the surgery with ultrasound guided technique with levobupivacaine 2.5mg/mL, 0.3mL/kg each side.
  The patient receives usual analgesia protocol.
  Interventions: Drug: Levobupivacaine Hydrochloride 2.5 MG/ML
- local infiltration of the trocar wounds (Active Comparator): local infiltration of the trocar wounds is realisated at the end of the surgery by the surgeon with levobupivacaine 2.5mg/mL 0.6mL/kg distributed in each trocar opening.
  The patient receives usual analgesia protocol.
  Interventions: Drug: Levobupivacaine Hydrochloride 2.5 MG/ML

INTERVENTIONS:
Drug: Levobupivacaine Hydrochloride 2.5 MG/ML — To compare TAP block versus local infiltration of the trocar wounds with levobupivacaine 2.5 mg/ml for post operative pain relief after laparoscopic appendicectomy in children

SUMMARY:
When performing laparoscopic appendectomy in children, regional anesthetic techniques are rou-tinely used concomitantly with general anesthesia. These techniques include local infiltration of the trocar wounds or transverse abdominal plane block (TAP block). In 2018, a position paper of the European Society of Pediatric Anaesthesiology advised for TAP block over local infiltration of the trocar wounds. However, there is no randomized study comparing both techniques in children. The aim of this study is to compare morphine consumption during the first 24 postoperative hours in children undergoing laparoscopic appendectomy and randomly allocated to either local infiltration of the trocar wounds or TAP block.

DETAILED DESCRIPTION:
This is a double blind randomized study with two parallel groups. Children between 3 and 15 years of age with indication of laparoscopic appendectomy will be approached for inclusion in this trial. Informed consent will be asked for from the parents and the child. Before surgery, patients will be randomized to either local infiltration of the trocar wounds or TAP block using sequentially numbered sealed envelope each with a random number inside. Patients with peritonitis will be excluded. A standardized analgesia protocol within the first 24 post-operative hours will be applied and the primary outcome is nalbuphine consumption during this time frame. Secondary outcomes include postoperative pain (FLACC assessment tool) and postoperative nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Age betwween 3 and 15 years
* Weight < or = 50 kg
* indicaction of coelioscopic appendicectomy
* ASA 1,2 or 3
* consent of the children and the holder of parental autority

Exclusion Criteria:

* Age<3 years or > 15years or weight > 50kg
* refusal of the children and the holder of parental autority
* ASA 4
* Peritonitis
* Patients with long term morphinic traitment
* Epilepsy
* Hepato-cellular insuffisiancy
* local anesthesia allergy or nalbuphine allergy
* coagulation abnomrmality
* exclusion of health insurance

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
cumulative dose of nalbuphine in the 24 first hours post surgery | 24 hours
  recording in mg/kg

SECONDARY OUTCOMES:
cumulative dose of nalbuphine H0-H12 post surgery | from beginning to 12th hour
  recording in mg/kg
cumulative dose of nalbuphine H13-H24 post surgery | From 13th hour to 24th hour
  recording in mg/kg
FLACC analgesia score at H1 H2 H6 H12 H24 | FLACC score will be performed from awakenig to 24 hours post surgery
  Face Leg Activity Cry Consolability heteroevaluation scale from 0 to 10
FLACC score mean | FLACC score will be performed from awakenig to 24 hours surgery
  Face Leg Activity Cry Consolability heteroevaluation scale from 0 to 10
individual variations of FLACC score | FLACC score will be performed from awakenig to 24 hours surgery
  Face Leg Activity Cry Consolability heteroevaluation scale from 0 to 10
timing of first injection of nalbuphine | in the first 24 post operative hours
  recording date and time of first injection
incidence of post operative nausea and vomiting | in the first 24 post operative hours
  recording the incidence post operative nausea and vomiting
timing of first standing up | in the first 24 post operative hours
  recording date and time of first standing up
adverse events | in the first 24 post operative hours
  adverse event monitoring

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Besancon, Besançon, France

IPD SHARING:
Plan to Share IPD: Undecided